CLINICAL TRIAL: NCT00279448
Title: Multicenter, Randomized, Open-Label Study To Compare The Efficacy, Tolerance And Quality Of Life Of 5 Years Of Adjuvant Exemestane (Aromasin) Therapy With 2.5 To 3 Years Of Adjuvant Tamoxifen Therapy, Followed By 2 To 2.5 Years Of Exemestane For A Total Duration Of 5 Years To Treat HR+ Post-Menopausal Patients With Non-Metastatic Breast Cancer
Brief Title: Exemestane As Treatment In Adjuvant For Post-Menopausal Patients With Non-Metastatic Breast Cancer
Acronym: TEAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EXEAPO-0028-118; A5991081
Record Dates: First submitted 2006-01-17; First posted 2006-01-19 (Estimated); Last update posted 2011-12-23 (Estimated); Status verified 2011-12

CONDITIONS: Breast Neoplasms
MeSH Terms: conditions — Breast Neoplasms | interventions — exemestane; Tamoxifen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental)
  Interventions: Drug: exemestane
- B (Active Comparator)
  Interventions: Drug: tamoxifen

INTERVENTIONS:
Drug: exemestane — On tablet of 25 mg per day during 5 years
  Other Names: Aromasin
  Arms: A
Drug: tamoxifen — Two tablets of tamoxifen 10 mg per day during 2.5 to 3 years followed by one tablet of exemestane 25 mg per day during 2 to 2.5 years for a total duration of 5 years of treatment
  Other Names: Kessar
  Arms: B

SUMMARY:
To compare recurrence free survival between two treatment groups (5 years with exemestane vs 2.5 to 3 years tamoxifen followed by 2 to 2.5 years of exemestane for a total duration of 5 years)

This Pfizer sponsored trial is part of an international collaboration of investigators conducting 7 similar yet independent studies in 9 countries. This study is designed to be part of the larger TEAM trial where the data from these 7 studies will be combined. A pre-specified analysis of the pooled data will be conducted. Link to TEAM Trial [971-ONC-0028-081/A5991026] Study Results: http://clinicaltrials.gov/ct2/show/results/NCT00036270?term=971-ONC-0028-081&rank=1

ELIGIBILITY:
Inclusion Criteria:

* HR+ post-menopausal patients with non-metastatic breast cancer

Exclusion Criteria:

* Any of the following: HR-, non-menopausal patient, metastatic breast cancer

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9779 (Actual)
Dates: Start 2002-01; Primary Completion 2008-11 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
To compare recurrence free survival between two treatment groups. | 2.75 years and 5 years

SECONDARY OUTCOMES:
The quality of life of patients treated with exemestane to that of patients treated with tamoxifen | Every 3 months during first year then every 6 months for 4 years
Overall survival between the 2 treatment groups | Every 3 months during first year then every 6 months for 4 years
Incidence of a second breast cancer (contralateral) between the 2 treatment groups | Every 3 months during first year then every 6 months for 4 years
General tolerance in the short- and long-term between the 2 treatment groups | Every 3 months during first year then every 6 months dor 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (54):
- France (54):
  - Pfizer Investigational Site, Marseille, Be1 01971
  - Pfizer Investigational Site, Compiègne, Be1 02256
  - Pfizer Investigational Site, Rennes, Be1 03677
  - Pfizer Investigational Site, Brest, Be1 04292
  - Pfizer Investigational Site, Aix-en-Provence
  - Pfizer Investigational Site, Amiens
  - Pfizer Investigational Site, Annecy
  - Pfizer Investigational Site, Avignon
  - Pfizer Investigational Site, Bayonne
  - Pfizer Investigational Site, Blois
  - Pfizer Investigational Site, Bordeaux
  - Pfizer Investigational Site, Brest
  - Pfizer Investigational Site, Cagne Sur Mer
  - Pfizer Investigational Site, Chalon-sur-Saône
  - Pfizer Investigational Site, Chaumont
  - Pfizer Investigational Site, Croix
  - Pfizer Investigational Site, Dijon
  - Pfizer Investigational Site, Douai
  - Pfizer Investigational Site, Draguignan
  - Pfizer Investigational Site, Dunkirk
  - Pfizer Investigational Site, Évreux
  - Pfizer Investigational Site, Hyres
  - Pfizer Investigational Site, L'Union
  - Pfizer Investigational Site, Le Havre
  - Pfizer Investigational Site, Lille
  - Pfizer Investigational Site, Lorient
  - Pfizer Investigational Site, Lyon
  - Pfizer Investigational Site, Mareuil-lès-Meaux
  - Pfizer Investigational Site, Marseille
  - Pfizer Investigational Site, Metz
  - Pfizer Investigational Site, Montauban
  - Pfizer Investigational Site, Montbéliard
  - Pfizer Investigational Site, Montélimar
  - Pfizer Investigational Site, Montpellier
  - Pfizer Investigational Site, Mougins
  - Pfizer Investigational Site, Nancy
  - Pfizer Investigational Site, Nantes
  - Pfizer Investigational Site, Neuilly
  - Pfizer Investigational Site, Nice
  - Pfizer Investigational Site, Nîmes
  - Pfizer Investigational Site, Paris
  - Pfizer Investigational Site, Pessac
  - Pfizer Investigational Site, Quincy-sous-Sénart
  - Pfizer Investigational Site, Reims
  - Pfizer Investigational Site, Ris-Orangis
  - Pfizer Investigational Site, Saint-Brieuc
  - Pfizer Investigational Site, Saint-Cloud
  - Pfizer Investigational Site, Saint-Herblain
  - Pfizer Investigational Site, Saint-Nazaire
  - Pfizer Investigational Site, Strasbourg
  - Pfizer Investigational Site, Toulon
  - Pfizer Investigational Site, Toulouse
  - Pfizer Investigational Site, Vandœuvre-lès-Nancy
  - Pfizer Investigational Site, Vannes

REFERENCES:
- [Derived] Leblanc A, Beltran-Bless AA, Pond GR, El Emam K, Juwara L, Clemons L, Bayani J, Pilgram L, Pharoah P, Mallon E, Taylor KJ, Markopoulos C, Dirix L, Vandermeer L, Hilton J, Savard MF, Bartlett JMS, Clemons M. Prognostic and predictive performance of PREDICT 2.1, PREDICT v3, and RSClin in node-negative early breast cancer: a TEAM pathology substudy. Breast Cancer Res Treat. 2026 Feb 5;215(3):74. doi: 10.1007/s10549-026-07909-5. PMID 41642493
- [Derived] Beltran-Bless AA, Pond GR, Bayani J, Barker SL, Spears M, Mallon E, Taylor KJ, Hasenburg A, Markopoulos C, Dirix L, Meershoek-Klein Kranenbarg E, van de Velde CJH, Rea DW, Vandermeer L, Hilton J, Bartlett JMS, Clemons M. Does RSClin provide additional information over classic clinico-pathologic scores (PREDICT 2.1, INFLUENCE 2.0, CTS5)? Breast. 2025 Oct;83:104528. doi: 10.1016/j.breast.2025.104528. Epub 2025 Jul 4. PMID 40633461
- [Derived] Bayani J, Kornaga EN, Crozier C, Jang GH, Bathurst L, Kalatskaya I, Trinh QM, Yao CQ, Livingstone J, Boutros PC, Spears M, McPherson JD, Stein LD, Rea D, Bartlett JMS. Identification of Distinct Prognostic Groups: Implications for Patient Selection to Targeted Therapies Among Anti-Endocrine Therapy-Resistant Early Breast Cancers. JCO Precis Oncol. 2019 Dec;3:1-13. doi: 10.1200/PO.18.00373. PMID 35100692
- [Derived] Derks MGM, Bastiaannet E, van de Water W, de Glas NA, Seynaeve C, Putter H, Nortier JWR, Rea D, Hasenburg A, Markopoulos C, Dirix LY, Portielje JEA, van de Velde CJH, Liefers GJ. Impact of age on breast cancer mortality and competing causes of death at 10 years follow-up in the adjuvant TEAM trial. Eur J Cancer. 2018 Aug;99:1-8. doi: 10.1016/j.ejca.2018.04.009. Epub 2018 Jun 6. PMID 29885375
- [Derived] Derks MGM, Blok EJ, Seynaeve C, Nortier JWR, Kranenbarg EM, Liefers GJ, Putter H, Kroep JR, Rea D, Hasenburg A, Markopoulos C, Paridaens R, Smeets JBE, Dirix LY, van de Velde CJH. Adjuvant tamoxifen and exemestane in women with postmenopausal early breast cancer (TEAM): 10-year follow-up of a multicentre, open-label, randomised, phase 3 trial. Lancet Oncol. 2017 Sep;18(9):1211-1220. doi: 10.1016/S1470-2045(17)30419-9. Epub 2017 Jul 18. PMID 28732650
- [Derived] Kalatskaya I, Trinh QM, Spears M, McPherson JD, Bartlett JMS, Stein L. ISOWN: accurate somatic mutation identification in the absence of normal tissue controls. Genome Med. 2017 Jun 29;9(1):59. doi: 10.1186/s13073-017-0446-9. PMID 28659176
- [Derived] Bartlett JM, Brookes CL, Piper T, van de Velde CJ, Stocken D, Lyttle N, Hasenburg A, Quintayo MA, Kieback DG, Putter H, Markopoulos C, Kranenbarg EM, Mallon EA, Dirix LY, Seynaeve C, Rea DW. Do type 1 receptor tyrosine kinases inform treatment choice? A prospectively planned analysis of the TEAM trial. Br J Cancer. 2013 Oct 29;109(9):2453-61. doi: 10.1038/bjc.2013.609. Epub 2013 Oct 3. PMID 24091623
- [Derived] van de Velde CJ, Rea D, Seynaeve C, Putter H, Hasenburg A, Vannetzel JM, Paridaens R, Markopoulos C, Hozumi Y, Hille ET, Kieback DG, Asmar L, Smeets J, Nortier JW, Hadji P, Bartlett JM, Jones SE. Adjuvant tamoxifen and exemestane in early breast cancer (TEAM): a randomised phase 3 trial. Lancet. 2011 Jan 22;377(9762):321-31. doi: 10.1016/S0140-6736(10)62312-4. PMID 21247627
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=EXEAPO-0028-118&StudyName=Exemestane%20As%20Treatment%20In%20Adjuvant%20For%20Post-Menopausal%20Patients%20With%20Non-Metastatic%20Breast%20Cancer
- See also: Link to TEAM Trial [971-ONC-0028-081/A5991026] Study Results — http://clinicaltrials.gov/ct2/show/results/NCT00036270?term=971-ONC-0028-081&rank=1